CLINICAL TRIAL: NCT03392376
Title: Agents Intervening Against Delirium in Intensive Care Unit (AID-ICU) A Randomized, Blinded, Placebo-controlled Trial
Brief Title: Agents Intervening Against Delirium in Intensive Care Unit
Acronym: AID-ICU
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zealand University Hospital (Other)
Collaborators: Centre for Research in Intensive Care (CRIC) (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); Scandinavian Critical Care Trials Group (Other); The Danish Centre of Applied Social Science (VIVE) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REG-169-2017
Record Dates: First submitted 2017-11-30; First posted 2018-01-08 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Delirium
Keywords: ICU Delirium; Haloperidol
MeSH Terms: conditions — Delirium | interventions — Haloperidol; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Haloperidol injection (Experimental): Haloperidol 2,5mg x 3 daily, with additional as needed doses to a maximum of 20mg/daily.
  Other name: Serenase
  Interventions: Drug: Haloperidol Injection
- Normal Saline (Placebo Comparator): Saline (0,9%)
  Interventions: Other: Saline (0,9%)

INTERVENTIONS:
Drug: Haloperidol Injection — ICU patients with diagnosed delirium are treated with 2,5mg haloperidol x 3 daily intravenously with additional as needed doses to a maximum of 20mg/daily.
  Other Names: Serenase
  Arms: Haloperidol injection
Other: Saline (0,9%) — ICU patients with diagnosed delirium are treated with 0,5ml isotonic saline x 3 daily and as needed doses to a maximum of 4ml/daily, corresponding to the algorithm in the experimental arm.
  Arms: Normal Saline

SUMMARY:
Delirium is a frequent condition in the Intensive Care Unit (ICU) with no existing evidence-based treatment. The aim of the AID-ICU study is to assess the benefits and harms of haloperidol treatment for the management of ICU acquired delirium.

DETAILED DESCRIPTION:
Delirium among critically ill patients in the intensive care unit (ICU) is a common condition associated with increased morbidity and mortality. No evidence-based treatment exist of this condition. Haloperidol is the most frequently used agent to treat ICU-related delirium, but according to the available literature there is no firm evidence of efficacy and safety of this intervention. AID-ICU aims to assess the benefits and harms of haloperidol in adult, critically ill patients with delirium in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Acute admission to the ICU AND
* Age ≥ 18 years AND
* Diagnosed delirium with validated screening Tool as either CAM-ICU or ICDSC

Exclusion Criteria:

* Contraindications to haloperidol
* Habitual treatment with any antipsychotic medication or treatment with antipsychotics in the ICU prior to inclusion
* Permanently incompetent (e.g. dementia, mental retardation)
* Delirium assessment non-applicable (coma or language barriers)
* Withdrawal from active therapy
* Fertile women (women < 50) with positive urine human chorionic gonadotropin (hCG) or plasma hCG.
* Consent according to national regulations not obtainable
* Patients under coercive measures by regulatory authorities
* Patients with alcohol-induced delirium (Delirium Tremens)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-06-13 (Actual); Primary Completion 2022-07-09 (Actual); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Days alive out of the hospital within 90 days post-randomization | 90 days
  Number of days alive and out of hospital
90-day mortality | 90 days
  Death from any cause within 90 days post-randomization
Hospital Length of Stay | 90 days
  Total number of days the patient is admitted to any hospital within the 90-day intervention period

SECONDARY OUTCOMES:
Number of days alive without delirium or coma in the ICU | Until ICU discharge, maximum 90 days
  Number of days where patients are both alive and free of delirium and coma
Number of patients with one or more serious adverse reactions to haloperidol and the total number of serious adverse reactions to haloperidol compared with placebo | Measured every day from inclusion until ICU discharge, maximum 90 days
  Serious adverse reactions are: Anaphylactic reactions, Agranulocytosis, Pancytopenia, Ventricular arrhythmia, Extrapyramidal symptoms, Tardive dyskinesia, Malignant Neuroleptic Syndrome, Acute hepatic failure
Usage of escape medicine | Measured every day from inclusion until ICU discharge, maximum 90 days
  Number of patients receiving escape medicine and number of days with escape medicine per patients
Number of days alive without mechanical ventilation within 90 days postrandomisation | Measured every day from inclusion until ICU discharge, maximum 90 days
  Number of days where patients are both alive and free of mechanical ventilation
Mortality | 1 year
  Landmark mortality 1 year post-randomisation
Quality of life (five level) | 1 year
  EQ-5D-5L total score 1 year post-randomisation (1-5 of each of the five domains)
Quality of life (overall self assessment) | 1 year
  EQ-Visual Analogue Scale 1 year post-randomisation (0-100)
Cognitive function 1 year after randomisation at selected sites | 1 year
  Repeated Battery for the Assesment of Neuropsychological Status score 1 year post-randomisation at selected sites (40-150)
Executive function 1 year after randomisation at selected sites | 1 year
  Trail Making Test 1 year post-randomisation at selected sites (40-150)
A health economic analysis | 90 days
  The analytic details will be based on the primary results of the trial (cost-benefit or cost-minimisation analyses)
Cognitive function at admission | At inclusion (within the first week)
  Informant Questionnaire on Cognitive Decline in the Elderly at ICU admission at selected sites (40-150)

CONTACTS AND LOCATIONS:
Overall Officials: OIe Mathiesen, MD, PhD, Study Chair — Zealand University Hospital; Anders Perner, MD,PhD, Study Chair — Rigshospitalet, Denmark; Jørn Wetterslev, MD, PhD, Study Chair — Copenhagen Trial Unit, Center for Clinical Intervention Research
Locations (16):
- Denmark (13):
  - Dept. Intensive Care, Aabenraa Hospital, Aabenraa
  - Dept. of Intensive Care, Aalborg University Hospital, Aalborg
  - Dept. of Intensive Care 4131, Copenhagen University Hospital, Rigshospitalet, Copenhagen
  - Dept. of Intensive Care, Herlev Hospital, Herlev
  - Dept. of Intensive Care, Herning Hospital, Herning
  - Dept. of Intensive Care, Nordsjaelland Hospital, Hillerød
  - Regionshospitalet Nordjylland, Hjørring, Hjørring
  - Dept. of Intensive Care, Holstebro Hospital, Holstebro
  - Dept. of Intensive Care, Zealand University Hospital, Køge, Køge
  - Dept. of Intensive Care, Nykøbing Falster Hospital, Nykøbing Falster
  - Dept of intensive care, Odense University Hospital, Odense
  - Dept. of Intensive Care, Zealand University Hospital Roskilde, Roskilde
  - Dept. of Intensive Care, Sønderborg Hospital, Sønderborg
- Dept. of Intensive Care, Helsinki University Central Hospital, Helsinki, Finland
- Dept. of Neurosurgical Intensive Care, San Gerardo Hospital, Monza., Monza, Italy
- UHW Adult Critical Care Cardiff, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mortensen CB, Andersen-Ranberg NC, Poulsen LM, Granholm A, Rasmussen BS, Kjaer MN, Lange T, Ebdrup BH, Collet MO, Andreasen AS, Bestle MH, Uslu B, Pedersen HS, Nielsen LG, Hastbacka J, Jensen TB, Damgaard K, Sommer T, Morgen M, Dey N, Citerio G, Estrup S, Egerod I, Samuelson K, Perner A, Mathiesen O. Long-term outcomes with haloperidol versus placebo in acutely admitted adult ICU patients with delirium. Intensive Care Med. 2024 Jan;50(1):103-113. doi: 10.1007/s00134-023-07282-7. Epub 2024 Jan 3. PMID 38170227
- [Derived] Andersen-Ranberg NC, Poulsen LM, Perner A, Wetterslev J, Estrup S, Hastbacka J, Morgan M, Citerio G, Caballero J, Lange T, Kjaer MN, Ebdrup BH, Engstrom J, Olsen MH, Oxenboll Collet M, Mortensen CB, Weber SO, Andreasen AS, Bestle MH, Uslu B, Scharling Pedersen H, Gramstrup Nielsen L, Toft Boesen HC, Jensen JV, Nebrich L, La Cour K, Laigaard J, Haurum C, Olesen MW, Overgaard-Steensen C, Westergaard B, Brand B, Kingo Vesterlund G, Thornberg Kyhnauv P, Mikkelsen VS, Hyttel-Sorensen S, de Haas I, Aagaard SR, Nielsen LO, Eriksen AS, Rasmussen BS, Brix H, Hildebrandt T, Schonemann-Lund M, Fjeldsoe-Nielsen H, Kuivalainen AM, Mathiesen O; AID-ICU Trial Group. Haloperidol for the Treatment of Delirium in ICU Patients. N Engl J Med. 2022 Dec 29;387(26):2425-2435. doi: 10.1056/NEJMoa2211868. Epub 2022 Oct 26. PMID 36286254
- See also: LINK to the AID-ICU webpage — http://www.cric.nu/aid-icu/